CLINICAL TRIAL: NCT04610385
Title: Comparative Study Between Ileal Conduit and Unilateral Cutaneous Ureterostomy With Separate Stomas Post Radical Cystectomy
Brief Title: Ileal Conduit Versus Cutaneous Ureterostomy After Radical Cystectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Hosam Mahdy, resident of urology, Assiut University
Other Study IDs: bladder caner treatment
Record Dates: First submitted 2020-08-28; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Patient Satisfaction; Bladder Cancer
MeSH Terms: conditions — Patient Satisfaction; Urinary Bladder Neoplasms | interventions — Cystectomy; Urinary Diversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ileal conduit
  Interventions: Procedure: radical cystectomy with urinary diversion
- cutaneous ureterostomy
  Interventions: Procedure: radical cystectomy with urinary diversion

INTERVENTIONS:
Procedure: radical cystectomy with urinary diversion — surgical removal of the urinary bladder and other organs and perform a urinary shunt

SUMMARY:
Bladder cancer is the most common malignancy of the urinary tract and accounts for about 3.2% of all cancer worldwide where it remains the seventh most commonly diagnosed malignancy in the male population. Causative risk factors can be broadly divided into inherited and acquired due to environmental exposure ,Tobacco smoking is the most important environmental risk factor for bladder cancer(1).

Histologically, over 90% of bladder tumors are transitional cell carcinomas. The other subtypes, such as squamous cell and adenocarcinoma, are uncommon and account for 5 and <2%, respectively(2).

Radical cystectomy with pelvic lymph node dissection with appropriate urinary diversion remains the mainstay of surgical treatment for muscle invasive bladder cancer and for high risk non muscle invasive disease. Select group of patients or those unfit or unwilling for surgery are managed by trimodal therapy utilizing transurethral resection and chemoradiotherapy.(3) The ideal urinary diversion should successfully preserve renal function while managing urinary outflow and minimizing morbidity to the patient(4).Several types of urinary diversion are present, continent and incontinent. Our study will focus on ileal conduit and cutaneous ureterostomy.

Although ileal conduit considered the standard method for incontinent urinary diversion, it is associated with early bowel related complications, i.e., bowel obstruction, prolonged ileus, and anastomotic leak which are mainly associated with bowel resection and anastomosis and late complications comprise ureteroenteric stricture, urinary fistula and stomal site complications in 25-60% of patients, including stomal stenosis, retraction, prolapsed, and parastomal herniation. Cutaneous ureterostomy may represent a method of choice for elderly and otherwise morbid patients due to its relative short duration and less bowel and metabolic complications but it has a high rate of stomal stenosis making perminant stenting is mandatory(5).

Cutaneous ureterostomy with separate stomas offers easy exchange of stents not need tertiary center with fluoroscopy or endescopy guidance compared to cutaneous ureterostomy with single stoma and this is preferable in our community.

ELIGIBILITY:
Inclusion Criteria:

* patients with bladder cancer eligible for surgery

Exclusion Criteria:

* Patients who refuse to contribute in this study.
* patients who are unfit for surgery.
* patients refusing cystectomy.
* patients with metastatic or inoperable cancer bladder

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bladder cancer eligible for radical cystectomy and will undergo either ileal conduit or unilateral cutaneous ureterostomy with separate stomas with age range from 45 to 85 years regardless of gender.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
quality of life measure | 1 year postoperative
  using FAST-BCI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsaturyan A, Sahakyan S, Muradyan A, Fanarjyan S, Tsaturyan A. A new modification of tubeless cutaneous ureterostomy following radical cystectomy. Int Urol Nephrol. 2019 Jun;51(6):959-967. doi: 10.1007/s11255-019-02145-x. Epub 2019 Apr 13. PMID 30982146
- [Background] Moeen AM, Safwat AS, Gadelmoula MM, Moeen SM, Abonnoor AEI, Abbas WM, ElGanainy EO, El-Taher AM. Health related quality of life after urinary diversion. Which technique is better? J Egypt Natl Canc Inst. 2018 Sep;30(3):93-97. doi: 10.1016/j.jnci.2018.08.001. Epub 2018 Aug 23. PMID 30145025
- [Background] Lee RK, Abol-Enein H, Artibani W, Bochner B, Dalbagni G, Daneshmand S, Fradet Y, Hautmann RE, Lee CT, Lerner SP, Pycha A, Sievert KD, Stenzl A, Thalmann G, Shariat SF. Urinary diversion after radical cystectomy for bladder cancer: options, patient selection, and outcomes. BJU Int. 2014 Jan;113(1):11-23. doi: 10.1111/bju.12121. PMID 24330062